CLINICAL TRIAL: NCT03386058
Title: Examining Carryover Effect in Patients Treated witH Spinal cOrd Stimulation (ECHO). An Open, Prospective, Multicenter Study.
Brief Title: Examining Carryover Effect in Patients Treated witH Spinal cOrd Stimulation (ECHO)
Acronym: ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); CHU de Quebec-Universite Laval (Other); Medisch Spectrum Twente (Other); Odense University Hospital (Other); Aalborg University Hospital (Other); Sahlgrenska University Hospital (Other); Diakoniekrankenhaus Friederikenstift (Other); Sunderby Hospital (Other); Erasmus Medical Center (Other); AZ Delta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SCS ECHO
Record Dates: First submitted 2017-12-06; First posted 2017-12-29 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2020-11

CONDITIONS: Neuralgia; Spinal Cord Stimulation
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: Open study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Temporary device deactivation
  Interventions: Device: Temporary device deactivation

INTERVENTIONS:
Device: Temporary device deactivation — Patient-controlled, temporary deactivation of implanted device

SUMMARY:
Spinal cord stimulation is a minimally invasive surgical treatment for severe, chronic, neuropathic pain that is refractory to conventional treatment.

The treatment consists of an electrode implanted in the epidural space of the spinal cord, either via a percutaneous approach (using the so-called percutaneous leads) or via a surgical (hemi-) laminectomy (using the so-called surgical leads or plate leads).

It is a well-known clinical observation that when activating or deactivating SCS stimulation, there is a variable interval before the patient perceives a clinical effect of the change. This variation goes by different names (carryover, echo, after effect, etc.) and might be dependent on the clinical condition and treatment duration. To our knowledge only very little research has been published on the topic of carryover effects; a recent study showed that the interval is highly variable between patients.

While patients may experience immediate pain relief at the onset of SCS treatment, the effect in patients with a long-term SCS treatment history may have different characteristics, possibly due to ongoing changes in the nervous system.

The aim of this pilot study is to lay the foundation for investigating the carryover effects in spinal cord stimulation.

This will be carried out in a mixed population of patients with different indications for SCS, and with different treatment durations.

Patients will be asked to deactivate their device via their remote control or with a magnet in a standardized fashion.

They will be asked to reactivate the device when specific parameters have been met, and the time is recorded.

DETAILED DESCRIPTION:
In the post-hoc analysis the carryover and reverse carryover effect will be analyzed and correlated to a number of parameters including, but not limited to: Indication, treatment duration, symptom duration, preoperative pain score, stimulation paradigm, gender, age.

Data will be collected and stored using a dedicated REDCap database under the auspices of Aarhus University.

ELIGIBILITY:
Inclusion Criteria:

* patient age minimum 18 years
* signed informed consent
* implanted with full SCS system for neuropathic pain
* SCS treatment duration minimum 6 months before inclusion
* maximum pain score 7 or less on a 0-10 NRS at the area of pain treated with SCS during the last 48 hours before study-related deactivation of the device

Exclusion Criteria

* any surgical SCS lead revision for the last 6 months before inclusion
* any changes in the programming patterns of the device (except patient-controlled changes in amplitude) for a minimum of 30 days before the study-related deactivation of the device
* any other ongoing neuromodulatory treatment (PNS, TENS, etc.)
* any other neuromodulatory treatment with lasting effect (RFA, sympathectomy, infiltration anesthesia, nerve blockade) within the last 60 days
* any changes in analgetic medication within the last 30 days (pn. dosings are allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Carryover/echo effect: Time from deactivation of device to cessation of treatment affect | Up to one week (may be repeated)
  Time from deactivation of device to cessation of treatment affect

SECONDARY OUTCOMES:
Reverse carryover/echo effect: Time from reactivation of device to full reestablishment of treatment effect | Up to one week (may be repeated)
  Time from reactivation of device to full reestablishment of treatment effect

CONTACTS AND LOCATIONS:
Overall Officials: Kaare Meier, MD PhD, Principal Investigator — Aarhus University Hospital
Locations (10):
- AZ Delta Roeselare/Menen/Torhout, Roeselare, Belgium
- CHU de Québec - Université Laval, Québec, Quebec, Canada
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense
- Diakovera Friederikenstift, Hanover, Germany
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Erasmus University Medical Center, Rotterdam
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Sunderby Hospital, Luleå

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolter T, Winkelmuller M. Continuous versus intermittent spinal cord stimulation: an analysis of factors influencing clinical efficacy. Neuromodulation. 2012 Jan-Feb;15(1):13-9; discussion 20. doi: 10.1111/j.1525-1403.2011.00410.x. Epub 2011 Dec 12. PMID 22151660
- [Background] Perruchoud C, Eldabe S, Batterham AM, Madzinga G, Brookes M, Durrer A, Rosato M, Bovet N, West S, Bovy M, Rutschmann B, Gulve A, Garner F, Buchser E. Analgesic efficacy of high-frequency spinal cord stimulation: a randomized double-blind placebo-controlled study. Neuromodulation. 2013 Jul-Aug;16(4):363-9; discussion 369. doi: 10.1111/ner.12027. Epub 2013 Feb 20. PMID 23425338
- [Derived] Meier K, de Vos CC, Bordeleau M, van der Tuin S, Billet B, Ruland T, Blichfeldt-Eckhardt MR, Winkelmuller M, Gulisano HA, Gatzinsky K, Knudsen AL, Hedemann Sorensen JC, Milidou I, Cottin SC. Examining the Duration of Carryover Effect in Patients With Chronic Pain Treated With Spinal Cord Stimulation (EChO Study): An Open, Interventional, Investigator-Initiated, International Multicenter Study. Neuromodulation. 2024 Jul;27(5):887-898. doi: 10.1016/j.neurom.2024.01.002. Epub 2024 Mar 7. PMID 38456888